CLINICAL TRIAL: NCT00779870
Title: Evaluating the Role of Oxidant/Anti-oxidant Balance and the Relationship of Asthma Severity on Airway Smooth Muscle Proliferation, Migration and Cytokine Release.
Brief Title: Airway Smooth Muscle and Asthma Severity
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Asthma UK (Other); Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Fan Chung, Professor, Imperial College London
Other Study IDs: 08/H0708/2
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Results first posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Asthma
Keywords: asthma severity; airway smooth muscle; oxidative stress
MeSH Terms: conditions — Asthma | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — endobronchial biopsies and cultured airway smooth muscle cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1: healthy volunteers
  Interventions: Other: bronchoscopy
- 2: mild asthmatics
  Interventions: Other: bronchoscopy
- 3: moderately-severe asthmatics
  Interventions: Other: bronchoscopy
- 4: severe asthmatics
  Interventions: Other: bronchoscopy

INTERVENTIONS:
Other: bronchoscopy — bronchoscopy under local anaesthetic and sedation to obtain endobronchial biopsies

SUMMARY:
Our hypothesis is that the severity of asthma is determined by the way in which airway smooth muscle cells grow and release inflammatory mediators. Our main objective is to establish how the properties of the airway smooth muscle cell varies with asthma severity. Environmental agents, such as cigarette smoke, and inflammation can give rise to oxidative stress - this is a process whereby harmful chemicals called free radicals are formed in the body and damage tissues. The damage caused can be limited/prevented by protective, or anti-oxidant mediators. We will also look at molecules involved in oxidative stress which may affect the way in which the airway smooth muscle grows and produces inflammatory mediators.

DETAILED DESCRIPTION:
Aims and Objectives The objective of this study is to examine whether the severity of asthma is related to (and possibly caused by) ASM dysfunction. Severe asthmatics have been shown to have more ASM in bronchial biopsies than non-severe asthmatics16. Because ASM cells can be obtained from bronchial biopsies obtained via bronchoscopy, we will examine endobronchial biopsies from mild, moderate and severe asthmatics, and healthy non-asthmatic subjects to compare features of remodelling (severe asthmatic subjects will have been assessed through the Difficult Asthma Protocol at the Royal Brompton Hospital24). In particular, we will focus on ASM mass, proliferation and changes in expression of different contractile proteins (α-actin and myosin) and chemokines, and will assess in vitro the response of ASM cells to stimulation by TGF-β and IL-1β. We will also examine the effect of dexamethasone on chemokine release and induced proliferation in vitro. We will also study enzymes and anti-oxidants involved in oxidative stress, such as Nox4, MnSOD and catalase, to look at their role in regulating ASM cell proliferation and chemokine synthesis. We want to see if there is an oxidant-anti oxidant balance in ASM in severe asthma compared to non-severe asthma.

AIM:

1. To establish the difference in ASM phenotype in asthma patients of differing severity of disease in terms of ASM mass, proliferation, migration and chemokine release.

Study design There will be 3 study visits. In the first two visits, the subjects will undergo spirometry with reversibility testing, a methacholine challenge test (to assess degree of bronchial hyper-responsiveness), skin prick tests and IgE levels (to assess atopic status), measurement of exhaled nitric oxide (as a non-invasive marker of inflammation), and the asthmatic subjects will complete an Asthma Control Questionnaire and an Asthma Quality of Life Questionnaire. The third visit will be on the day admission for the bronchoscopy.

Study protocol:

Visit 1 - screening visit

* Explain purpose of study- address any queries/concerns
* History and examination
* Skin prick tests
* Blood test for full blood count, clotting profile and IgE
* Measurement of exhaled nitric oxide (eNO)
* Spirometry pre and post β agonist
* Completion of Asthma Control Questionnaire and
* Completion of Asthma Quality of Life Questionnaire

Visit 2 - Methacholine challenge test

Visit 3 - Day admission for fibreoptic bronchoscopy

ELIGIBILITY:
Inclusion criteria - Asthma Age 18-60 Physician diagnosis of asthma Intermittent/mild, moderate and severe asthma as per GINA guidelines [1]

For the severe asthma subjects, they will also have the following:

Major characteristics (at least one of the following criteria)

* Treatment with continuous or near continuous (>50% of year) oral corticosteroids
* Requirement for treatment with high dose inhaled corticosteroids (ICS) Minor characteristics (at least 2 out of the following)

  1. Requirement for daily treatment with a controller medication in addition to ICS e.g. LABA, theophylline, leukotriene antagonist
  2. Asthma symptoms requiring SABA on a daily or near daily basis
  3. Persistent airways obstruction (FEV1 <80% predicted, diurnal PEF variation >20%)
  4. One or more emergency care visits for asthma per year
  5. 3 or more steroid "bursts" per year
  6. Prompt deterioration with ≤ 25% reduction in oral or ICS
  7. Near fatal asthma event in the past

     Reference [1] GINA - The Global Initiative for Asthma. www.ginasthma.com

     Exclusion criteria - Asthma Intubation for asthma within 6 months of entry into this study Current smokers, or less than 3 years since quitting smoking (< 5 pack/years) Less than 4 weeks from an exacerbation On steroid-sparing agent or immunosuppressant such as azathioprine, methotrexate and ciclosporin Concomitant anti-IgE therapy On anti-platelet or anti-coagulant drugs Low platelet count Pregnancy or breast-feeding Previous bronchoscopy within three months of this study

     Healthy volunteer subjects:

     We are aiming for 5 atopic and 5 non-atopic healthy volunteers.

     Inclusion criteria:

     Age 18 - 60 Non smokers (or less than 5 pack/yrs if ex-smokers) Normal lung function

     Exclusion criteria:

     History of asthma or allergic rhinitis Any chronic illness Current smokers, or less than 3 years since quitting smoking (< 5 pack/years) PC20 less than 16mg/ml On anti-platelet or anti-coagulant drugs Low platelet count Pregnancy or breast-feeding Previous bronchoscopy within three months of this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Mild, moderate and severe asthmatics, with a control group of healthy non-smoking volunteers
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kian F Chung, MBBS MD FRCP DSc, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Michaeloudes C, Chang PJ, Petrou M, Chung KF. Transforming growth factor-beta and nuclear factor E2-related factor 2 regulate antioxidant responses in airway smooth muscle cells: role in asthma. Am J Respir Crit Care Med. 2011 Oct 15;184(8):894-903. doi: 10.1164/rccm.201011-1780OC. PMID 21799075

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Results of the low number of participants the mild and moderate asthma patients were combined to Non severe group
Groups:
- Healthy: Healthy Participant
- Non-severe Asthma: Patients with mild and moderate asthma
- Severe Asthma: Patients with severe asthma
Period: Overall Study
Arm/Group | Healthy | Non-severe Asthma | Severe Asthma
Started | 5 | 6 | 7
Completed | 5 | 6 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy | Non-severe Asthma | Severe Asthma | Total
Number analyzed (Participants) | 5 | 6 | 7 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.67 (6.3) | 38.17 (8.5) | 36.67 (4.12) | 36.5 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Missing data from participant
  Participants
    number analyzed (Participants) | 3 | 6 | 6 | 15
    Female | 1 | 1 | 2 | 4
    Male | 2 | 5 | 4 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 5 | 6 | 7 | 18

OUTCOME MEASURES:

1. Primary Outcome: Difference in ASM Mass Between Groups
Time Frame: at time of bronchoscopy, an average of 1 hour
Population: No data collected
Arm/Group | Healthy | Non-severe Asthma | Severe Asthma
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Difference in ASM Proliferation, Migration and Cytokine Release Between Groups
Time Frame: at time of bronchoscopy, an average of 1 hour
Population: Data not collected
Arm/Group | Healthy | Non-severe Asthma | Severe Asthma
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Difference in Intracellular Oxidative Stress Mechanisms From ASM Between Groups
Description: Expression of Nrf2 protein
Time Frame: at time of bronchoscopy, an average of 1 hour
Measure: Mean (Full Range); unit: relative expression unit
Arm/Group | Healthy | Non-severe Asthma | Severe Asthma
Number analyzed (Participants) | 5 | 6 | 7
relative expression unit | 2 [1.1 to 2.4] | 3 [1.1 to 3.6] | 3 [1.2 to 4.2]
Statistical Analysis 1: Comparison: Healthy vs Non-severe Asthma; Test type: Superiority; p = 0.06, t-test, 2 sided
Statistical Analysis 2: Comparison: Healthy vs Severe Asthma; Test type: Superiority; p = 0.8, t-test, 2 sided

4. Secondary Outcome: Correlation Between ASM Mass and Airway Hyper-responsiveness (PC20)
Time Frame: at the time of bronchoscopy, an average of 1 hour
Population: No data collected
Arm/Group | Healthy | Non-severe Asthma | Severe Asthma
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Healthy | Non-severe Asthma | Severe Asthma
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes